CLINICAL TRIAL: NCT05239000
Title: Pilot Randomized Clinical Trial of Geriatric Comanagement or Geriatric Guided Supportive Care for Older Patients With Head and Neck Cancer Receiving Radiation and Chemotherapy
Brief Title: A Study Comparing Geriatric Co-Management With Geriatric Guided Supportive Care in Older Patients Receiving Chemoradiation Therapy for Their Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-016
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer
Keywords: Supportive Care; Older Patients with Head and Neck Cancer Receiving Radiation and Chemotherapy; 22-016
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: The study design is a randomized pilot clinical trial with two arms. Enrolled patients are those aged ≥70 years with newly diagnosed or post-operative head and neck squamous cell carcinoma. Patients will be undergoing radiation with concurrent chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- geriatric co-management (Experimental): Geriatric co-management involves a consultation with a geriatrician prior to initiating head and neck radiation and chemotherapy. Consultation with geriatricians can occur in-person or remotely via telemedicine. During this visit, the geriatrician will review the results of the eRFA and create a plan to manage geriatric deficits. Geriatric co-management involves optimization of comorbid conditions, management of polypharmacy, and supportive care referrals to address geriatric deficits. Geriatricians also work in conjunction with the treating oncologists to ensure patients have appropriate pain management and bowel regimens. Additional follow up visits after the initial consultation are at the discretion of the geriatrician may vary between patients depending on the clinical need.
  Interventions: Other: geriatric co-management
- geriatric guided supportive care (Experimental): Geriatric guided supportive care will be carried out by oncologists. After the patient completes the eRFA, an automated report is generated that identifies the patient's geriatric deficits. The automated report also includes suggested interventions for each deficit (e.g, referral to physical therapy. For instance, automated suggestions for a patient with a history of falls include consultation with physical therapy, neurologic evaluation, a home safety evaluation, or use of supportive devices. Automated recommendations for patient with high level of distress or depression include referral to psychiatry or social work, involvement in a cancer support group, or additional time spent addressing questions and fears. The oncology team will review the automated report from the eRFA and create an intervention plan prior to initiation of head and neck radiation and chemotherapy.
  Interventions: Other: geriatric guided supportive care

INTERVENTIONS:
Other: geriatric co-management — Geriatric co-management involves a consultation with a geriatrician prior to initiating head and neck radiation and chemotherapy.
  Arms: geriatric co-management
Other: geriatric guided supportive care — Geriatric guided supportive care will be carried out by oncologists. After the patient completes the eRFA, an automated report is generated that identifies the patient's geriatric deficits.
  Arms: geriatric guided supportive care

SUMMARY:
The researchers are doing this study to see whether geriatric co-management or geriatric guided supportive care are good approaches for managing side effects in older patients who have head and neck cancer and are receiving chemoradiation therapy. This study will provide valuable information about different ways to manage side effects in older patients receiving chemoradiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65
* Pathologically (histologically or cytologically) diagnosis of head and neck cancer of oral cavity, oropharynx, larynx, or hypopharynx
* Patient will receive a 6 to 7 week course of intensity modulated radiation therapy and concurrent chemotherapy either in definitive or post-operative setting
* Able to read and understand English
* Able to provide informed consent

Exclusion Criteria:

* Patients who have previously consulted with or are followed by a geriatrician
* Inability to use telemedicine if unable to present to clinic visits in person
* Inability to complete the eRFA (patient is unable to comprehend or answer questions included on the eRFA)
* Treatment with proton therapy
* Patients on therapeutic clinical trials of experimental therapies or those not receiving standard of care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
proportion of patients with hospital admission (geriatric co-management arm) | 2 years
  The proportion of patients hospitalized during the course of chemoradiation either at MSKCC or an outside hospital will be assessed for each arm.
proportion of patients with hospital admission (geriatric guided supportive care arm) | 2 years
  The proportion of patients hospitalized during the course of chemoradiation either at MSKCC or an outside hospital will be assessed for each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm